CLINICAL TRIAL: NCT01495130
Title: Mechanically-Manipulated Transrectal Ultrasound (TRUS) During Robotic-Assisted Laparoscopic Prostatectomy (RALP)
Brief Title: Transrectal Ultrasound (TRUS) in Finding Tumors During Robotic-Assisted Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4P-10-9; NCI-2011-03570 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-11-29; First posted 2011-12-19 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (TRUS) (Experimental): Patients undergo TRUS during RALP.
  Interventions: Procedure: ultrasound imaging; Procedure: robot-assisted laparoscopic surgery

INTERVENTIONS:
Procedure: ultrasound imaging — Undergo transrectal ultrasound
  Other Names: ultrasonography; ultrasound; ultrasound test
Procedure: robot-assisted laparoscopic surgery — Undergo robotic-assisted laparoscopic prostatectomy

SUMMARY:
This pilot clinical trial studies mechanically-manipulated ultrasound in finding tumors during robotic-assisted surgery in patients with prostate cancer. Diagnostic procedures, such as ultrasound, may help find prostate cancer and find out how far the disease has spread during surgery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To assess the feasibility and limitations of using a mechanically-manipulated transrectal ultrasound (TRUS) probe for TRUS evaluation during a da Vinci robotic-assisted laparoscopic prostatectomy (RALP). II. To collect TRUS evaluation data during RALP to guide us in deciding whether and how the mechanical manipulation of the TRUS probe will allow sufficient clarity of ultrasound imaging. OUTLINE: Patients undergo TRUS during RALP. After the completion of study treatment, patients are followed up at 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Robotic Assisted Laparoscopic Prostatectomy

Exclusion Criteria:

* Known or discovered rectal pathology
* Bleeding hemorrhoids
* Rectal stenosis
* Any prior rectal surgeries
* Prior rectal radiation
* Any known rectal disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of patients who have negative margins when a TRUS probe is used during RALP procedure without introducing additional complications. | 7 days post-RALP

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Ukimura, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States